CLINICAL TRIAL: NCT05938283
Title: Pilot Study of Hypertrophic Cardiomyopathy & Implantable Cardioverter Defibrillator Assessment: (Subcutaneous vs Transvenous)
Acronym: HICD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Boston Scientific Corporation (Industry); Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 158953
Record Dates: First submitted 2023-06-13; First posted 2023-07-10 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Implantable Defibrillator User; Hypertrophic Cardiomyopathy; Implantable Cardioverter Ventricular Lead Dysfunction or Complication; Ventricular Arrythmia
Keywords: Transvenous Implantable Defibrillator; Subcutaneous Implantable Defibrillator
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Defibrillators, Implantable

STUDY DESIGN:
Intervention Model Description: Pilot randomised control trial, randomised 1:1 for Transvenous: Subcutaneous
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transvenous Implantable Defibrillator (Active Comparator): Routine TV ICD implant
  Interventions: Device: Implantable Cardioverter Defibrillator implant
- Subcutaneous Implantable Defibrillator (Active Comparator): SICD ICD implant as per study protocol
  Interventions: Device: Implantable Cardioverter Defibrillator implant

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator implant — ICD implant to protect patients from life threatening ventricular tachycardia or ventricular fibrillation

SUMMARY:
Pilot randomised trial to assess recruitment for a larger trial to compare the efficacy and adverse effects of the subcutaneous and transvenous ICD in patients with hypertrophic cardiomyopathy (HCM) and indication for ICD therapy, with no requirement for pacing

DETAILED DESCRIPTION:
This study aims to test the feasibility of conducting a trial to investigate the use of subcutaneous implantable defibrillator (SICD) in patients with hypertrophic cardiomyopathy (HCM) and to determine whether SICD produces more complications than conventional, transvenous implantable defibrillator (TV ICD).

The primary analysis for the main trial is designed to test whether the S-ICD is non-inferior to the TV-ICD with respect to the primary endpoint of inappropriate shock treatment and complications. For the incidence of the primary endpoint statistical significance and 99% confidence intervals are calculated using Cox' proportional hazards model. Non-inferiority is considered to be established if the upper boundary of the one-sided 99% confidence interval did not exceed 1.92 (absolute difference < 12%).

Participant duration is expected to be 14 months. (12 months follow up post device implant) Recruitment duration expected to be 6-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Hypertrophic Cardiomyopathy and a referred for ICD therapy with no pacing requirement.

Exclusion Criteria:

* Patients with sustained ventricular tachycardia less than 170 bpm
* Patients having an indication for pacing therapy. E.g. sick sinus syndrome.
* Patients failing appropriate QRS/T-wave sensing with the automated S-ICD ECG automated patient screening provided by Boston Scientific
* A minimum of 1 sensing vector passing in supine, standing.
* Patients with incessant ventricular tachycardia
* Patients who have had a previous ICD implant
* Patient who receives cardiac contractility modulation therapy or are likely to receive cardiac contractility modulation therapy
* Patients with a serious known concomitant disease with a life expectancy of less than one year
* Patients with circumstances that prevent follow-up (no permanent home or address, transient, etc.)
* Patients who are unable to give informed consent
* Patients who are not suitable for TV-ICD implantation, according to the discretion of the physician, are not screened for enrolment (SVC occlusion).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Rate of recruitment | through study completion, expected at 10 months to 1 year
  Assessment of rate of recruitment per month
Composite of inappropriate shock and ICD related complications | 12 months
  Rate of inappropriate shocks and ICD related complications across the patients over a 12 month period.

SECONDARY OUTCOMES:
All- cause mortality | 12 months
  % of patients who die
MACE events | 12 months
  Major Adverse Cardiac Event (MACE), defined as cardiac death, myocardial infarction, percutaneous coronary intervention, coronary artery bypass grafting and/or any valve surgery.
Appropriate shocks and patients with appropriate shocks | 12 months
  Rate over 12 months determined by IBHRE accredited Cardiac Scientist
Inappropriate shocks and patients with inappropriate shocks | 12 months
  Rate over 12 months determined by IBHRE accredited Cardiac Scientist
Complications | 12 months
  individually, defined as infections, bleedings, thrombotic events, pneumothorax, perforation/tamponade, lead reposition and lead- or device failures
Cardiac decompensation | 12 months
  Measured by admissions for Heart failure or unplanned outpatient appointments.
Crossovers to the other arm | 12 months
  Amount of patients moving from SICD to TV group and visa versa over 12 month period.
Appropriate shock treatment in ATP or monitor zone | 12 months
  Rate over 12 months determined by IBHRE accredited Cardiac Scientist
Quality of life assessed by SF-36 survey | 12 months
  Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high QOL.
Quality of life assessed by EQ5D survey | 12 months
  Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high QOL.
Cardiac (pre-) syncope events | 12 months
  rate of patients with these events over a 12 month period
Time to successful therapy | 12 months
  Time in months or days from implant to date of succesful therapy
First shock conversion efficacy | 12 months
  % of first shocks that cardiovert ventricular arrhythmia
Implant procedure time | Procedure duration- average of 2 hours expected
  Duration of implant from needle to skin to skin closure.
Hospitalization rate | 12 months
  Rate of patient hospitalisation for cardiac and non-cardiac causes over a 12 month period.
Fluoroscopy time | Procedure duration- average of 2 hours expected
  Amount of fluoroscopy required to complete implant procedure, expected fluoroscopy time of approximately 1 minute per patient.

OTHER OUTCOMES:
Drop out rate | 12 months
  % of patients that do not complete the sudy
Data Quality | 12 months
  % of data completed
Eligibility of SICD | 12 months
  % Of patients referred for recruitment was SICD screening making patients illegible. Either Yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided